CLINICAL TRIAL: NCT02751502
Title: Home Based Adaptive Arm Training for Children With Hemiplegia
Brief Title: Home Based Adaptive Arm Training for Children
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of enrollment and funding + Covid-19 pandemic
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-01326
Record Dates: First submitted 2016-04-19; First posted 2016-04-26 (Estimated); Results first posted 2022-02-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Hemiplegia
Keywords: Children; Pediatrics; Arm; Upper limb; bimanual training; physical training
MeSH Terms: conditions — Hemiplegia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Bimanual-to-unimanual device home training program (Experimental)
  Interventions: Device: m2 Bimanual Arm Trainer (BAT)
- Conventional non-device home training program (No Intervention): Subjects receive 6 weeks of ongoing usual and customary care schedule of home physical and occupational therapy as usual and customary care independent of the study.

INTERVENTIONS:
Device: m2 Bimanual Arm Trainer (BAT) — Patients in the device group will be asked to train specific movements repeatedly with the device for 45 minutes five days a week for 6 weeks and compliance will be monitored through training logs and remotely
  Arms: Bimanual-to-unimanual device home training program

SUMMARY:
Twenty pediatric patients aged 5-17 years with Acquired Brain Injuries (ABI) will be randomized to receive either a bimanual-to-unimanual device home training program (10 subjects) or a conventional non-device home training program (10 subjects) for a period of 6 weeks.

The specific aims of this proposal are to:

Aim 1: Introduce home-based targeted upper limb training in children with hemiplegia from ABI (Acquired Brain Injuries) using a bimanual-to-unimanual training approach It is hypothesized that child-friendly home-based upper limb bimanual-to-unimanual training will lead to greater compliance and improved motor outcome on the Fugl Myer Scale compared to a conventional home training program.

Aim 2: Improve the understanding of the pattern of recovery of isolated joint movements in the pediatric population with hemiplegia following ABI.

It is hypothesized that individuals receiving device-based bimanual-to-unimanual training will show improvement in active range of motion across upper limb joints compared with a conventional home training program.

ELIGIBILITY:
Inclusion Criteria:

* Acquired Brain Injury at least 3 months prior to enrollment.
* Unilateral hemiparesis
* History of compliance with home exercise programs in the past.

Exclusion Criteria:

* Any social or medical problem that precludes compliance with the protocol
* Comorbid seizure disorder or other neurological disease
* Treatment with botulinum toxin or intrathecal baclofen in the 3 months preceding enrollment
* Implanted neuromodulatory or electronic device or other complicating illness
* Lack of capacity to consent

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2017-01; Primary Completion 2021-02-09 (Actual); Study Completion 2021-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renat Sukhov, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University Langone Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Whole Population: Data reported under one arm, as randomization into arms has not occurred yet.
Period: Overall Study
Arm/Group | Whole Population
Started | 4
Completed | 0
Not Completed | 4
Not completed — Lack of funding | 4

BASELINE CHARACTERISTICS:
Arm/Group | Whole Population
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Quality of Bimanual Hand Measured by Fugl-Meyer Scale
Description: Measure of impairments in motor functioning and recovery in children post hemiplegia.
Time Frame: 6 Weeks
Population: Study terminated prior to complete data collection
Arm/Group | Whole Population
Number analyzed (Participants) | 0

2. Primary Outcome: Change From Baseline in Timed Performance of Standardized Manual Activities Measured by Hand Assessment Test
Time Frame: 6 Weeks
Population: Study terminated prior to complete data collection
Arm/Group | Whole Population
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Study terminated prior to complete data collection.
Arm/Group | Whole Population
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-25): https://cdn.clinicaltrials.gov/large-docs/02/NCT02751502/Prot_SAP_000.pdf